CLINICAL TRIAL: NCT05625308
Title: Effect of Natural Compounds on the Severity of HPV-induced Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV-NAT-COM
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Papilloma; Cervix Lesion
MeSH Terms: conditions — Papilloma | interventions — epigallocatechin gallate; Folic Acid; Vitamin B 12; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: 40 HPV-positive women displaying chronic cervicitis, mild dysplasia or moderate dysplasia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-treatment with EGCG, FA, B12, and HA (Experimental): One tablet per day containing 200 mg of EGCG, 400 mcg of Folic Acid, 1 mg of Vitamin B12 and 50 mg of Hyaluronic Acid for twelve weeks.
  Interventions: Dietary Supplement: Epigallocatechin gallate, Folic acid, Vitamin B12, and Hyaluronic Acid
- Control (No Intervention): Untreated women.

INTERVENTIONS:
Dietary Supplement: Epigallocatechin gallate, Folic acid, Vitamin B12, and Hyaluronic Acid — One tablet per day containing 200 mg of EGCG, 400 mcg of Folic Acid, 1 mg of Vitamin B12 and 50 mg of Hyaluronic Acid.
  Arms: Co-treatment with EGCG, FA, B12, and HA

SUMMARY:
To test the efficacy of a newly-commercialized formula, 40 HPV-positive women displaying chronic cervicitis, mild dysplasia or moderate dysplasia. Women in the study group took one tablet per day containing 200 mg of EGCG, 400 mcg of Folic Acid, 1 mg of Vitamin B12 and 50 mg of Hyaluronic Acid for twelve weeks. Women in the control group received no treatment.

ELIGIBILITY:
Inclusion Criteria:

* HPV infections
* Occurrence of low-grade cervical lesions

Exclusion Criteria:

* Diagnosis of malignancy or severe cervical lesions
* Concurrent uterine pathologies
* Pregnancy or intended to seek pregnancy in the next three months
* Cancer

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Regression of cervical lesions | 12 weeks
  The actual outcome was to measure the rate of regression of the lesions, from moderate to mild, from mild to none.

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Aragona, MD, Principal Investigator — Clinica Alma Res
Locations (1):
- Clinica Alma Res, Roma, Italy

IPD SHARING:
Plan to Share IPD: No